CLINICAL TRIAL: NCT07260565
Title: Impact of a Sequential Isokinetic Fatigue Protocol Followed by Ankle Strengthening After Botulinum Toxin Injection Into Spastic Plantar Flexors on Foot Lift Strength and Walking
Acronym: ISOTOX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Victor Pauchet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-A00591-48; 2025-A00591-48 (Other: ID-RCB)
Record Dates: First submitted 2025-09-25; First posted 2025-12-03 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Spasticity of the Plantar Flexors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard rehabilitation protocol (Other): Patients in this groupe will undergo a standard rehabilitation programme five times a week, Monday to Friday, combining physiotherapy and adapted physical activity.
  Interventions: Procedure: standard rehabilitation programme
- isokinetic rehabilitation protocol (Experimental): Patients in this group will undergo isokinetic rehabilitation five times a week, Monday to Friday, and will receive treatment combining physiotherapy, adapted physical activity (see standard rehabilitation protocol) and strengthening on an isokinetic dynamometer.
  Interventions: Procedure: Isokinetic rehabilitation protocol.

INTERVENTIONS:
Procedure: Isokinetic rehabilitation protocol. — Patients in group will undergo isokinetic rehabilitation therapy five times a week, Monday to Friday, combining physiotherapy, adapted physical activity (see standard rehabilitation protocol) and strengthening exercises on an isokinetic dynamometer.
  Arms: isokinetic rehabilitation protocol
Procedure: standard rehabilitation programme — Patients in group will undergo a standard rehabilitation programme five times a week, Monday to Friday, combining physiotherapy and adapted physical activity.
  Arms: standard rehabilitation protocol

SUMMARY:
Spastic foot drop (speed- and force-dependent hypertonia) is one of the most common neuro-orthopaedic disorders following brain injury. It has a negative impact on walking and is closely linked to independence in activities of daily living.

This disorder combines a deficit in muscle strength in the plantar flexors and extensors with pathological hypertonia of the plantar flexors, causing an imbalance in ankle flexion and resulting in equinus deformity of the foot.

Botulinum toxin is the first-line pharmacological treatment for focal spasticity of neurological origin, and its effectiveness is directly linked to the quality and quantity of associated rehabilitation care. However, the associated rehabilitation protocols remain vague and are based on general recommendations combining: stretching of muscles and tendons, muscle strengthening of spastic muscles, their agonists and antagonists, and functional work. The standard rehabilitation protocol used in our centre will be detailed in the study protocol.

The isokinetic dynamometer is an open-chain muscle strengthening tool that has the advantage of introducing a concept of reproducible assessment and rehabilitation.

This reproducibility is difficult to guarantee with the rehabilitation techniques practised by a therapist, whose applied force and precision may vary from one session to another. We have therefore developed a sequential muscle strengthening protocol combining strengthening work - fatigue of the triceps surae followed by muscle strengthening work of the foot lifters.

The aim of this work is to determine the effects of this protocol compared to conventional rehabilitation aimed at promoting the post-injection effects of botulinum toxin.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient with spastic hemiplegia (regardless of cause)
* MAS 1-2 spasticity of the plantar flexors
* Deficit of the foot lifters at the minimum stage of contraction with movement
* Patient who has received botulinum toxin injections in the plantar flexors
* Patient who has been informed about the research and has given their written and signed informed consent
* Patient affiliated with a social security scheme or beneficiary of such a scheme

Exclusion Criteria:

* Refusal of consent
* Patient with severe cognitive impairment (MMSE <23/30)
* Surgery on the affected lower limb
* Patient unable to read, write or understand French
* Patient who is pregnant or breastfeeding, in accordance with Article L1121-5 of the CSP
* Vulnerable patients according to Article L1121-6 of the CSP
* Adult patients under guardianship, curatorship or judicial protection
* Patients unable to give their consent in person according to Article L.1121-8 of the CSP or adults protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Strength of the foot lifters | At the baseline, and after 1 month of rehabilitation course
  The strength of the foot lifters will be assessed by the maximum peak torque of the foot lifters at 60° (rPT 60°) measured using an isokinetic dynamometer. The primary endpoint is the change in rPT 60° between the value at inclusion and the value at the end of rehabilitation. This endpoint will be compared between the two arms.

SECONDARY OUTCOMES:
rPT values | At the baseline, after 1 month of rehabilitation course , after 3 month follow-up and after 6 month follow-up
  rPT values
Peak torque resistance | At the baseline, after 1 month of rehabilitation course, after 3 month follow-up and after 6 month follow-up
  Measured using an isokinetic dynamometer at different angular velocities.
Measurement of the agonist/antagonist ratio | At the baseline, after 1 month of rehabilitation course , after 3 month follow-up and after 6 month follow-up
  using the isokinetic dynamometer at different visits.
The spasticity score measured | Before the rehabilitation protocol, during the consultation for the botulinum toxin injection , after 1 month of rehabilitation course , after 3 month follow-up and after 6 month follow-up
  using the Modified Aschworth Scale and stretch reflex measurement at different visits.
The distance covered during a 6-minute walk test and the walking speed measured during a 10-metre walk test at the various follow-up visits. | Before the rehabilitation protocol, during the consultation for the botulinum toxin injection, after 1 month of rehabilitation course, after 3 month follow-up and after 6 month follow-up
  The distance covered during a 6-minute walk test and the walking speed measured during a 10-metre walk test at the various follow-up visits.
The exercise tolerance score | Before the rehabilitation protocol, during the consultation for the botulinum toxin injection, after 1 month of rehabilitation course , after 3 month follow-up and after 6 month follow-up
  Using the Borg scale
Clinical improvement in spasticity, | After 3 month follow-up and after 6 month follow-up
  which will be assessed by the doctor in charge of the patient
Collect the number of adverse events | At the baseline, before the rehabilitation protocol, after 1 month of rehabilitation course, after 3 month follow-up and after 6 month follow-up
  Collect the number of adverse events

IPD SHARING:
Plan to Share IPD: Undecided